CLINICAL TRIAL: NCT01644656
Title: Non-invasive Diagnosis of Portal Hypertension by Acoustic Radiation Force Impulse (ARFI) Imaging of the Liver and Spleen in Patients With Chronic Liver Disease
Brief Title: Non-invasive Diagnosis of Portal Hypertension With Acoustic Radiation Force Impulse (ARFI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01582
Record Dates: First submitted 2012-06-19; First posted 2012-07-19 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Portal Hypertension; Chronic Liver Disease
Keywords: portal hypertension; cirrhosis; ARFI; diagnostic study
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Disease | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acoustic radiation force impulse (ARFI) (Experimental): Imaging of liver and spleen using modified ultrasound
  Interventions: Device: ARFI ultrasound

INTERVENTIONS:
Device: ARFI ultrasound — ARFI imaging of the liver and spleen will be performed immediately before transjugular liver biopsy and HVPG procedures
  Other Names: acoustic radiation force impulse

SUMMARY:
The aim of this diagnostic study is to evaluate the efficacy of ARFI imaging (a specific type of ultrasound) in assessing the pressure of the portal vein (the major vein passing through the liver) and the amount of liver fibrosis in patients with chronic liver disease.

DETAILED DESCRIPTION:
DESIGN The study is designed as a prospective, cross-sectional, diagnostic study in which the investigators will evaluate the use of ARFI to diagnose clinically significant portal hypertension (CSPH defined as hepatic veous pressure gradient (HVPG)greater than 10 mmHg), taking HVPG measurements as gold standard.

METHODOLOGY

* The study will be performed at the VA Connecticut Healthcare System-West Haven and Yale.
* Study population will be recruited among patients from the VA/Yale Liver Clinics or outside hospitals that are referred to VA/Yale for a transjugular liver biopsy and hepatic venous pressure gradient measurement as part of their routine care.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85 years
* compensated chronic liver disease with suspected or confirmed liver cirrhosis sent for transjugular liver biopsy as part of their routine care
* signed informed consent

Exclusion Criteria:

* known contraindications to the performance of an HVPG measurement or a trans-jugular biopsy
* portal thrombosis
* previous surgical or transjugular portosystemic shunt
* previous total or partial splenectomy
* presence of comorbid conditions conferring a life expectancy of less than 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-07; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
correlation of acoustic radiation force impulse (ARFI) measurement of organ stiffness with hepatic venous pressure gradient (HVPG) | Both outcome measurements (ARFI measurements and HVPG) will be obtained within an average time frame of 4-8 hours
  Both measurements are estimates of portal hypertension (defined as equal to HVPG greater than 10 mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia-Tsao, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (2):
- United States (2):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut